CLINICAL TRIAL: NCT02453945
Title: Use of a Support Bra to Reduce Pain and Improve Surgical Healing in Women Undergoing Sternotomy for Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Medbuy Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R.E.B. number: 15-144
Record Dates: First submitted 2015-02-19; First posted 2015-05-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pain; Disruption or Dehiscence of Closure of Sternum or Sternotomy; Quality of Life
Keywords: pain; comfort; healing; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Support Bra (Experimental): ClearPoint Medical Support Bra worn by patients during their post-cardiac surgery hospital stay (approximately 5-7days).
  Interventions: Device: Adjustable Support Bra
- Control (No Intervention): Usual Care

INTERVENTIONS:
Device: Adjustable Support Bra — A ClearPoint Medical support bra
  Arms: Medical Support Bra

SUMMARY:
The primary purpose of this study is to examine whether a properly fitted support bra on females improves their quality of life post-sternotomy. Specifically, does a support bra reduce discomfort, pain and wound dehiscence.

DETAILED DESCRIPTION:
Participants will be randomized to one arm of the study. One group will be fitted for a support bra and will be asked to wear this bra 24 hours a day for their 6 week post-course. They will submit to 3 questionnaires (at hospital discharge, at 3 weeks post-op and at their 6 week post-op visit with their surgeon. They will diary over this 6 week period re: pain, comfort, wound healing. The group in the no bra arm will also be measured for breast size and will submit to 3 questionnaires (at the same intervals) and will be asked to diary over their 6 week post-op course re: pain, comfort, wound healing. Chronic pain and quality of life markers will be assessed through a 6month and 1 year follow-up telephone call and questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 yrs) who are undergoing cardiac surgery with a sternotomy

Exclusion Criteria:

* Patients who have had a previous mastectomy
* Previous radiotherapy to the chest
* Patients who do not read, write or have issues comprehending English
* Patients with cognitive impairments who will not be able to comply with the research study protocol
* Patients requiring physical restraints
* Patients requiring the application of a sternal binder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analog Scale | Post-operative period (approximately 5-7days),
  Patients will be tracked post-operatively during their hospital stay (approximately 5-7days), at their 6 week follow up visit, 6-months and 1-year after their surgery date.
Pain - Visual Analog Scale | 6 weeks
  6-week post-op visit
Pain - Pt questionnaire | 6 months after surgery
Pain - Patient questionnaire | 1 year after surgery

SECONDARY OUTCOMES:
Comfort - Patient Questionaires | Post-operative period in hospital (approximately 5-7days)
  Patients will be tracked post-operatively during their hospital stay (approximately 5-7days), at their 6 week follow up visit, 6-months and 1-year after their surgery date.
Comfort - Patient Questionaires | 6-week post-op visit
  Patients will be tracked post-operatively during their hospital stay (approximately 5-7days), at their 6 week follow up visit, 6-months and 1-year after their surgery date.
Comfort - Patient Questionaires | 6-months
  Patients will be tracked post-operatively during their hospital stay (approximately 5-7days), at their 6 week follow up visit, 6-months and 1-year after their surgery date.
Comfort - Patient Questionaires | 1-year
  Patients will be tracked post-operatively during their hospital stay (approximately 5-7days), at their 6 week follow up visit, 6-months and 1-year after their surgery date.
Sternal Wound Dehiscence - Medical Documentation in chart | In hospital post-operative period (approximately 5-7days).
  Patients will be tracked during their hospital stay (approximately 5-7days) for sternal wound complications.
Quality of life pre cardiac surgery - Lawton ADL (Activity of daily living) scale | Pre-op
  Patients will be assessed pre-op, at 6-months after surgery and again at the 1 year point.
Quality of life pre cardiac surgery - SF12 | Pre-op
  Patients will be assessed pre-op, at 6-months after surgery and again at the 1 year point.
Quality of life post cardiac surgery - Lawton ADL (Activity of daily living) scale | 6 months
Quality of life post cardiac surgery - SF12 | 6 months
Quality of life post cardiac surgery - Lawton ADL (activity of daily living) scale | 1 year
Quality of life post cardiac surgery - SF12 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St Michael, Toronto, Ontario, Canada